CLINICAL TRIAL: NCT03951714
Title: 12-wks Randomised Controlled Trial to Explore the Effect of a Smartphone App. Connected to an Add-on Device System Fitted on pMDI Inhaler on Adherence to Medications Intake and Clinical Outcomes in Difficult-to-treat Asthmatic Patients
Brief Title: Effect of the Use of an add-on Device Connected to a Smartphone App on Difficult-to-treat Asthmatic Patient's Adherence
Acronym: ADVICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CLI-01535AA1-01
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Asthma
Keywords: Post-market study
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Reference (Other): Control experience using marketed application to record medication intake without reminders from the app
  Interventions: Behavioral: Marketed experience application on adherence
- Intervention (Experimental): Full experience using marketed application, with all functionalities enabled
  Interventions: Behavioral: Marketed experience application on adherence

INTERVENTIONS:
Behavioral: Marketed experience application on adherence — To evaluate the effect of electronic capture of medication intake through a smartphone app on treatment's adherence

SUMMARY:
The purpose of this Study is to assess the effect of a smartphone application connected to an add-on device system fitted on Pressured Metered Dose Inhaler (PMDI) on adherence to take medications as prescribed and clinical outcomes in difficult-to-treat asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written informed consent obtained prior to any study-related procedures
* Male or female patient aged 18 years and above
* Patient with established diagnosis of asthma for at least 6 months
* Patient on maintenance therapy (Fixed dose combination ICS/LABA) with high dose of ICS
* Patient with ACT score <20 at screening and at randomization
* Non- or ex-smoker who smoked ≤ 10 Pack-years prior to screening
* Patient must have their own Android® or iPhone operating system (IOS) smartphone
* Ability to use the pMDI device correctly

Exclusion Criteria:

* Patient with an asthma exacerbation or respiratory tract infection requiring systemic steroids and/or antibiotics within 1 to 3 month prior to screening
* Patient with a history of near-fatal asthma
* Clinically relevant and uncontrolled cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, psychiatric or any other disorder that would put the safety of the subject at risk through participation, or which would affect the analysis
* Patient not able to be compliant with the study requirements.
* Patient with a BMI > 40
* Patient working on night shifts
* Patient participating in the clinical phase of an interventional trial or have done so within the last 30 days prior to screening.
* Patient who has an already planned major surgery or hospitalization
* Female patient who is pregnant or lactating or who plans to become pregnant in the next 4 months.
* Patient with a history of hypersensitivity to any of the components of Foster pMDI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in adherence rate to entire treatment period | From baseline to end of participation (up to 3 months)
  Adherence Rate of doses correctly taken twice daily

OTHER OUTCOMES:
Asthma Control Test score | From baseline to end of participation (up to 3 months)
  Change from Baseline
Test of the Adherence to Inhalers score | From baseline to end of participation (up to 3 months)
  Change from Baseline
Percentage of days without intake of rescue medication | From baseline to end of participation (up to 3 months)
  Change from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Annaliese Linnhoff, Principal Investigator — Research Center for Medical Studies Praxis für Lungen- und Bronchialheilkunde
Locations (1):
- Barlow Medical Centre, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614
- See also: Structured Summary Data Results on Chiesi Clinical Study Register — https://www.chiesi.com/en/chiesi-clinical-study-register/